CLINICAL TRIAL: NCT05919407
Title: IMproving Symptomatic Treatment With Pyridostigmine and Amifampridine: a Randomized Double-blinded, Placebo Controlled Crossover Trial in Patients With Myasthenia Gravis (IMPACT-MG)
Brief Title: Pyridostigmine and Amifampridine for Myasthenia Gravis
Acronym: IMPACT-MG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: NMD Pharma A/S (Industry)
Responsible Party: Principal Investigator, Martijn R. Tannemaat, MD PhD, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL78666.058.21
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Pyridostigmine Bromide; Amifampridine; Alkalies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pyridostigmine (Experimental): The dose of pyridostigmine will be based on the patient's prior experience with pyridostigmine under the assumption that the patient already gained sufficient experience during their disease course to know which dose is effective for them as patients are advised by their treating neurologist to continually adjust their dose based on their symptoms and side effects.
  Interventions: Drug: Pyridostigmine
- Placebo (pyridostigmine) (Placebo Comparator): Same as "Experimental", however capsules contain placebo.
  Interventions: Drug: Placebo
- Amifampridine (base) with modified release (Experimental): Patients will receive amifampridine 2 dd 15 mg and amifampridine 2 dd 30 mg as add-on to the pre-study dose of pyridostigmine.
  Interventions: Drug: Amifampridine (base) with modified release
- Placebo (amifampridine) (Placebo Comparator): Same as "Experimental", however capsules contain placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Participants will receive pyridostigmine 10 mg tablets.
  Arms: Pyridostigmine
Drug: Amifampridine (base) with modified release — Participants will receive amifampridine (base) with modified release 15 mg or 30 mg tablets.
  Arms: Amifampridine (base) with modified release
Drug: Placebo — The placebo tablets will be identical apart from the active substance (pyridostigmine)
  Arms: Placebo (pyridostigmine)
Drug: Placebo — The placebo tablets will be identical apart from the active substance (amifampridine base)
  Arms: Placebo (amifampridine)

SUMMARY:
A randomized, double-blind, placebo controlled, crossover intervention study evaluating the effect of pyridostigmine (part 1) and amifampridine (part 2) in Myasthenia Gravis (MG).

DETAILED DESCRIPTION:
In the first part of the study, patients who are currently using pyridostigmine will be randomly allocated to one of two consecutive treatment periods in which patients either first receive placebo and then their usual dose of pyridostigmine, or vice versa. Each treatment period lasts 5 days with a 2-day wash-out period between each treatment period. Measurements will be performed at every last day of a treatment period (day 5 and day 12).

In the second part of the study the effect of two doses of amifampridine as add-on to pyridostigmine will be studied. Patients will be randomly assigned to either one of three treatment sequences; 1) amifampridine 30 mg - amifampridine 60 mg - placebo or 2) amifampridine 60 mg - placebo - amifampridine 30 mg or 3) placebo - amifampridine 30 mg - amifampridine 60 mg. Again, each treatment period consists of 5 days and will be separated by a 2-day wash-out period. Measurements will be performed at every last day of treatment (day 19, day 26 and day 33).

Patients will have the option to participate in a substudy to characterize the pharmacokinetics (PK) and pharmacodynamics (PD) of amifampridine in AChR positive MG patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. AChR positive myasthenia gravis (ocular or generalized)
3. Current use of pyridostigmine
4. MGFA Clinical Classification I-IV
5. Receiving a stable dose of MG treatment (other than pyridostigmine). If applicable:

   1. A stable steroid regimen for 1 month
   2. Nonsteroidal immunosuppressants: i. Azathioprine, mycophenolate mofetil, cyclosporine or other nonsteroid immunosuppressive agents start > 3 months ago and a stable regimen for 1 month. ii. Rituximab start > 6 months ago, complement inhibitors and Fc receptor inhibitors start > 6 months ago and a stable regimen for 3 months.

Additional inclusion criteria for part 2 To be eligible for participation in part 2 of the study patients must score >10 points on the MGII questionnaire at inclusion.

We will include a maximum of 5 patients with a MGFA class I (i.e. 20 percent of the total number of included patients) to ensure that this study accurately reflects the clinical population.

Exclusion Criteria:

1. Use of intravenous immunoglobulin or plasma exchange <4 weeks or planned during the trial.
2. Thymectomy < 6 months, or thymectomy (expected) to take place during the trial
3. Use of other acetylcholinesterase inhibitors than pyridostigmine
4. Pregnancy, lactation or intention to become pregnant during the study
5. Treatment with amifampridine is contraindicated. Contraindications include a history of epilepsy, uncontrolled asthma, inherited QT syndrome / a prolonged QT interval (as indicated by ECG), any drug known to cause QT c-prolongation, any drug known to lower the epileptic threshold, a known hypersensitivity reaction to the active substance or to any of the excipients.
6. The patient is unable to fill out the study questionnaires or be interviewed in Dutch, or is unable to undergo the tests needed for the study, or is unable to give informed consent for participation in the study.
7. The investigator can exclude patients for this trial which are deemed not suitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-09-22 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
A clinically relevant change in Myasthenia Gravis Impairment Index (MGII) compared to placebo. | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),

SECONDARY OUTCOMES:
Change on 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) compared to placebo | Assessed on Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),
Change on the 15-item revised version of the Myasthenia Gravis Quality of Life questionnaire (MG-QoL15r) compared to placebo | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),
A clinically relevant change (≥2 points change) on the Myasthenia Gravis Activities of Daily Living (MG-ADL) score compared to placebo. | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),
A clinically relevant change (≥3 points change) on the Quantitative Myasthenia Gravis (QMG) score compared to placebo. | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),
Number of patients not able to complete first wash-out period due to an increase in myasthenic symptoms. | Assessed on Day 1 (crossover)
Number of times escape medication is used (including effect on symptoms) | Assessed on Day 1, Day 5 and Day 12 (cross-over),
Trough concentrations of pyridostigmine and amifampridine | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33 (cross-over),
Peak Plasma Concentration (Cmax) | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Area under the concentration-time curve (AUC0-8) | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Time of maximum concentration (Tmax) | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Serum half-life (T1/2) | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Trough concentration (Ctrough) | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Dose-response between serum concentrations of amifampridine and hand grip strength as measured with hand-held dynamometer. | Assessed on Day 19, Day 26 and Day 33 (cross-over),
Utility as assessed by the 5-level EQ-5D (EQ-5D-5L) | Assessed on Day 1, Day 5, Day 12, Day 19, Day 26 and Day 33
Healthcare use as assessed by the adapted iMCQ (iMTA Medical Consumption Questionnaire) | Assessed on Day 1
  The iMCQ is adapted by omitting the modules on medication and travel. The recall period for the iMCQ is set to 12 months.
Productivity as assessed by the adapted iPCQ (iMTA Productivity Cost Questionnaire) | Assessed on Day 1
  The recall period for the iPCQ is set to 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands